CLINICAL TRIAL: NCT02846376
Title: Phase I Study of Single-agent and Combined Checkpoint Inhibition After Allogeneic Hematopoietic Stem Cell Transplantation in Patients at High Risk for Post-transplant Recurrence
Brief Title: Single Agent and Combined Inhibition After Allogeneic Stem Cell Transplant
Acronym: CPIT-002
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2016-0526
Record Dates: First submitted 2016-06-24; First posted 2016-07-27 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia and Myelodysplastic Syndrome
MeSH Terms: conditions — GATA2 Deficiency | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to Groups A, and B in a 1:1 fashion. If the safety endpoint is met for each of these groups, enrollment to Group C will open. Each patient will be monitored for toxicities for at least 28 days before the next patient is added to the same cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - Nivolumab (Experimental): Nivolumab for 12 doses, on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34
  * Dose level 1: 1 mg/kg
  * Dose level 2: 3 mg/kg
  Interventions: Drug: Nivolumab
- Group B - Ipilimumab (Experimental): Ipilimumab for 6 doses on day 1 of weeks 1, 4, 7, 10, 13, 16
  * Dose level 1: 0.3 mg/kg
  * Dose level 2: 1.0 mg/kg
  * Dose level 3: 3.0 mg/kg
  Interventions: Drug: Ipilimumab
- Group C - Nivolumab + Ipilimumab (Experimental): * Nivolumab 3 mg/kg for 12 doses, on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34
  * Ipilimumab for 6 doses on day 1 of weeks 1, 4, 7, 10, 13, 16
    * Dose level 1: 0.3 mg/kg
    * Dose level 2: 0.6 mg/kg
    * Dose level 3: 1.0 mg/kg
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a fully humanized immunoglobulin 4 (IgG4) monoclonal antibody (mAb) which binds to PD-1 (CD279) with nanomolar affinity and shows a high degree of specificity for PD-1; blocking binding of PD-1 to PD-L1 and PD-L2. Nivolumab binds selectively to human PD-1 and does not bind to other members of the cluster of differentiation protein 28 (CD28) family.
  Other Names: Bristol-Myers Squibb (BMS-936558)
  Arms: Group A - Nivolumab; Group C - Nivolumab + Ipilimumab
Drug: Ipilimumab — Ipilimumab is a recombinant, human mAb that binds to the cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4). Ipilimumab is an immunoglobulin 1 (IgG1) kappa immunoglobulin with an approximate molecular weight of 148 kilo-Daltons (kDa). Ipilimumab is produced in mammalian (Chinese hamster ovary) cell culture.
  Other Names: BMS-734016
  Arms: Group B - Ipilimumab; Group C - Nivolumab + Ipilimumab

SUMMARY:
The purpose of the study is to determine the safety and benefit of nivolumab, ipilimumab or the combination of nivolumab with ipilimumab given after bone marrow transplant for patients with acute myelogenous leukemia and myelodysplastic syndrome.

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To assess the safety of single-agent and combined checkpoint inhibition with nivolumab and ipilimumab in patients with acute myelogenous leukemia and myelodysplastic syndrome who have undergone hematopoietic stem cell transplantation and are at high risk for post-transplant recurrence.
* Safety endpoint: The composite endpoint consisting of the occurrence of at least one treatment-related limiting toxicity (after checkpoint inhibitor treatment is initiated) defined as a ≥ grade 4 non-hematologic toxicity as specified by the CTCAE. Exceptions listed in section 5.9 apply to this endpoint as well. If 3 of 7 patients in a single cohort experience a treatment-related limiting toxicity, that single cohort will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and local guidelines.
2. Be 18 years or older and 70 years or younger on the day of signing consent
3. Have a confirmed diagnosis of non-M3 acute myeloid leukemia (AML) (Intermediate-II is high risk. Our population will consist of Intermediate-II and high risk patients or any FLT3+ AML) or IPSS intermediate -2 or high risk myelodysplastic syndrome (MDS) (Appendices A and B).
4. Have an available 6/6 related donor or an unrelated donor with a 10/10 match for HLA-A, B, C, DRB1 and DQ antigen who consents to provide a marrow or peripheral blood stem cell allograft. Typing is by DNA techniques: intermediate resolution for A, B and C, and high resolution for DRB1/DQ
5. Be receiving one of the following conditioning regimen: fludarabine at a dose of 30 mg/m2 IV daily for 5 days, busulfan at a dose of 130 mg/m2 IV daily for 2 days, and rabbit antithymocyte globulin (ATG) at a dose of 2 mg/kg IV daily for 2 days OR fludarabine at a dose of 30 mg/m2 IV daily for 4 days, melphalan at a dose of 140 mg/m2 for one day with or without ATG at a dose of 2 mg/kg IV daily for 2 days
6. Be deemed eligible for an allogenic stem cell transplantation as per institutional guidelines of the Blood and Marrow Transplantation Program at John Theurer Cancer Center at Hackensack University Medical Center
7. Patients with adequate organ function as measured by:

   * Cardiac: left ventricular ejection fraction at rest > 50%
   * Hepatic: serum total bilirubin < 1.5x upper limit of normal for age as per local laboratory (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome); ALT and AST < 4x upper limit of normal for age as per local laboratory
   * Renal: serum creatinine < 2x upper limit of normal for age (as per local laboratory). For patients with serum creatinine above the normal range, a glomerular filtration rate (measured as per institutional practice, typically creatinine clearance) equal to or greater than 60 mL/min (corrected to 1.73m2 body surface area) is required.
   * Pulmonary: FEVl, FVC and DLCO (corrected for Hb) >50% predicted.
8. Have a performance status of 2 or lower on ECOG performance scale.
9. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

   Version 1.0 23Mar2017 Page 4 of 73
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should agree to ongoing pregnancy testing, to be performed prior to each dosing of ipilimumab and nivolumab. See Note below for definition of WOCBP.
11. Women must not be breastfeeding.
12. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab, and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product, even if they have had a vasectomy. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception). See Note below for definition of WOCBP.
13. Females of childbearing potential must be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years. See Note below for definition of WOCBP.

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 20 mg/day prednisone equivalents) for at least 4 weeks prior to study drug administration. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 20 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
2. Is unable or unwilling to sign informed consent.
3. Has an active, known, or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
4. Patients should be excluded if they have a condition such as GVHD requiring systemic treatment with either corticosteroids (> 20 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 20 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalation corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 20 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
5. As there is potential for hepatictoxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
6. Has received a prior allogeneic stem cell transplant.
7. Has a history of hypersensitivity to nivolumab, ipilimumab, or any of its excipients, or severe hypersensitivity reaction to any previous monoclonal antibody.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Day 1 of checkpoint inhibitor treatment administration or who has not recovered (i.e., t administration mAb) within 4 weeks prior to t dose of trial treatment. Rituximab within that time frame is allowed.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Note: Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 20 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring intravenous systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known acquired immunodeficiency syndrome (AIDS).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has the presence of a large accumulation of ascites or pleural effusions, which would be a contraindication to the administration of methotrexate for GVHD prophylaxis.
19. Has known history of grade 3 or 4 GVHD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Safety: The occurrence of at least one treatment-related limiting toxicity defined as a ≥ grade 4 non-hematologic toxicity as specified by the CTCAE 4.0. | After treatment is initiated through 100 days of discontinuation of dosing.
  Exceptions are: Isolated Grade 4 amylase or lipase values that are not associated with symptoms or clinical manifestations of pancreatitis and decrease to < Grade 4 within 1 week of onset and isolated Grade 4 electrolyte imbalances/abnormalities that are not associated with clinical sequelae and are corrected with supplementation/appropriate management within 72 hours of their onset. If 3 of 7 patients in a single cohort experience a treatment-related limiting toxicity, that single cohort will be terminated.

SECONDARY OUTCOMES:
Toxicities: Common Terminology Criteria for Adverse Events (CTCAE) will be used for the assessment and grading of all toxicities experienced by patients enrolled into this study. | Through 100 days of discontinuation of dosing.
  Patients will be assigned to Groups A, B, and C in a 1:1:1 fashion. Each patient will be monitored for toxicities for at least 14 days before the next patient is added to the same cohort. The toxicity will be evaluated for all adverse events with grade 3 or grade 4 observed in each cohort and presented as counts (proportion).
Assessment of blood immune reconstitution by sequencing to determine diversity and highest frequency clonal specificities | At consent for subjects and within 30 days pre allo transplant conditioning for donors, at apheresis, and day 1 of week 1 of protocol treatment (tx) and then weeks 4,7,12,18,26, and at 9,12,15,18 mos post-transplant and at relapse if within 18 mos of tx.
Tumor site immune phenotyping | If bone marrow biopsy is available prior to allogeneic transplantation conditioning and then at time of relapse within 18 months following initiation of therapy.
  Absolute number of PD-L1/L2-bearing activated helper T cell subpopulations from bone marrow biopsy will be examined for two time points prior to conditioning and time of progression (within 18 months post-checkpoint inhibitor initiation) using Poisson regression analysis with GEE described in analysis of blood phenotype above.
Assessment of complete response (CR) rate | Assess at 3, 6 and 12 months after transplant
  The estimates of the CR will be presented as count (proportion) and corresponding exact binomial 95% confidence intervals for proportion at each time point.
Assessment of blood phenotype | At consent for subjects and within 30 days pre allogeneic transplant conditioning for donors, at apheresis, and day 1 of week 1 of protocol tx and weeks 4,7,12,18,26, and at 9,12,15,18 months post-transplant and at relapse if within 18 months of tx.
  Phenotype analysis of for T cells, Dendritic cells, Macrophages, Myeloid derived suppressor cells, B cells, natural killer (NK) cells, natural killer T (NKT) cells, Plasma Cytokine levels: Multiplex 25 Cytokine - Luminex via Flow Cytometric Phenotype Analysis
Assessment of blood TCR repertoire via TCR Immunoseq Assay Profiling | At consent for subjects and within 30 days pre allogeneic transplant conditioning for donors, at apheresis, and day 1 of week 1 of protocol tx and weeks 4,7,12,18,26, and at 9,12,15,18 months post-transplant and at relapse if within 18 months of tx.
  Via TCR Immunoseq for T cell receptor Vbeta complementarity determining region CDR3 highest frequency specificities.
Assess tumor site TCR repertoire using Poisson regression analysis with generalized estimating equations (GEE) | When bone marrow biopsy is available prior to allogeneic transplantation conditioning and then at time of relapse within 18 months following initiation of therapy.
  GEE method will be performed by utilizing the Statistical Analysis Software (SAS 9.4) procedure (PROC) generalized linear product analysis (GENMOD) with Poisson distribution, log link function and independent covariance structure.
Assess tumor site PD-L1/2 expression | When bone marrow biopsy is available prior to allogeneic transplantation conditioning and then at time of relapse within 18 months following initiation of therapy.
  If viable biopsy material is unavailable for research purposes, Dr. Korngold's lab will access fixed archival tumor materials for preparing tumor lysates and possibly for retrieving T cell DNA for repertoire analysis.
Efficacy as assessed by progression free survival (PFS) | At 12 months after treatment is initiated
  PFS is defined as time interval from date of protocol treatment initiation to pathologic disease progression or death from any cause. PFS will be estimated using Kaplan-Meier method and probabilities will be calculated for 12 months.
Efficacy as assessed by progression free survival (PFS) | At 18 months after treatment is initiated
  PFS is defined as time interval from date of protocol treatment initiation to pathologic disease progression or death from any cause. PFS will be estimated using Kaplan-Meier method and probabilities will be calculated for 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pecora, MD, Principal Investigator — Hackensack UMC; James McCloskey, MD, Principal Investigator — Hackensack UMC; Jamie Koprivnikar, MD, Principal Investigator — Hackensack UMC
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin S, Baldock SC, Ghoneim AT, Child JA. Defective neutrophil function and microbicidal mechanisms in the myelodysplastic disorders. J Clin Pathol. 1983 Oct;36(10):1120-8. doi: 10.1136/jcp.36.10.1120. PMID 6311878
- [Background] Martino R, Iacobelli S, Brand R, Jansen T, van Biezen A, Finke J, Bacigalupo A, Beelen D, Reiffers J, Devergie A, Alessandrino E, Mufti GJ, Barge R, Sierra J, Ruutu T, Boogaerts M, Falda M, Jouet JP, Niederwieser D, de Witte T; Myelodysplastic Syndrome subcommittee of the Chronic Leukemia Working Party of the European Blood and Marrow Transplantation Group. Retrospective comparison of reduced-intensity conditioning and conventional high-dose conditioning for allogeneic hematopoietic stem cell transplantation using HLA-identical sibling donors in myelodysplastic syndromes. Blood. 2006 Aug 1;108(3):836-46. doi: 10.1182/blood-2005-11-4503. Epub 2006 Apr 4. PMID 16597592
- [Background] Fukuda T, Hackman RC, Guthrie KA, Sandmaier BM, Boeckh M, Maris MB, Maloney DG, Deeg HJ, Martin PJ, Storb RF, Madtes DK. Risks and outcomes of idiopathic pneumonia syndrome after nonmyeloablative and conventional conditioning regimens for allogeneic hematopoietic stem cell transplantation. Blood. 2003 Oct 15;102(8):2777-85. doi: 10.1182/blood-2003-05-1597. Epub 2003 Jul 10. PMID 12855568
- [Background] Diaconescu R, Flowers CR, Storer B, Sorror ML, Maris MB, Maloney DG, Sandmaier BM, Storb R. Morbidity and mortality with nonmyeloablative compared with myeloablative conditioning before hematopoietic cell transplantation from HLA-matched related donors. Blood. 2004 Sep 1;104(5):1550-8. doi: 10.1182/blood-2004-03-0804. Epub 2004 May 18. PMID 15150081
- [Background] de Lima M, Anagnostopoulos A, Munsell M, Shahjahan M, Ueno N, Ippoliti C, Andersson BS, Gajewski J, Couriel D, Cortes J, Donato M, Neumann J, Champlin R, Giralt S. Nonablative versus reduced-intensity conditioning regimens in the treatment of acute myeloid leukemia and high-risk myelodysplastic syndrome: dose is relevant for long-term disease control after allogeneic hematopoietic stem cell transplantation. Blood. 2004 Aug 1;104(3):865-72. doi: 10.1182/blood-2003-11-3750. Epub 2004 Apr 15. PMID 15090449
- [Background] Armand P, Nagler A, Weller EA, Devine SM, Avigan DE, Chen YB, Kaminski MS, Holland HK, Winter JN, Mason JR, Fay JW, Rizzieri DA, Hosing CM, Ball ED, Uberti JP, Lazarus HM, Mapara MY, Gregory SA, Timmerman JM, Andorsky D, Or R, Waller EK, Rotem-Yehudar R, Gordon LI. Disabling immune tolerance by programmed death-1 blockade with pidilizumab after autologous hematopoietic stem-cell transplantation for diffuse large B-cell lymphoma: results of an international phase II trial. J Clin Oncol. 2013 Nov 20;31(33):4199-206. doi: 10.1200/JCO.2012.48.3685. Epub 2013 Oct 14. PMID 24127452
- [Background] Ansell SM, Lesokhin AM, Borrello I, Halwani A, Scott EC, Gutierrez M, Schuster SJ, Millenson MM, Cattry D, Freeman GJ, Rodig SJ, Chapuy B, Ligon AH, Zhu L, Grosso JF, Kim SY, Timmerman JM, Shipp MA, Armand P. PD-1 blockade with nivolumab in relapsed or refractory Hodgkin's lymphoma. N Engl J Med. 2015 Jan 22;372(4):311-9. doi: 10.1056/NEJMoa1411087. Epub 2014 Dec 6. PMID 25482239
- [Background] Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer--preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010 Oct;37(5):430-9. doi: 10.1053/j.seminoncol.2010.09.005. PMID 21074057
- [Background] O'Day SJ, Hamid O, Urba WJ. Targeting cytotoxic T-lymphocyte antigen-4 (CTLA-4): a novel strategy for the treatment of melanoma and other malignancies. Cancer. 2007 Dec 15;110(12):2614-27. doi: 10.1002/cncr.23086. PMID 18000991
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Fong L, Small EJ. Anti-cytotoxic T-lymphocyte antigen-4 antibody: the first in an emerging class of immunomodulatory antibodies for cancer treatment. J Clin Oncol. 2008 Nov 10;26(32):5275-83. doi: 10.1200/JCO.2008.17.8954. Epub 2008 Oct 6. PMID 18838703
- [Background] Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor D, Salama AK, Taylor M, Ott PA, Rollin LM, Horak C, Gagnier P, Wolchok JD, Hodi FS. Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17. doi: 10.1056/NEJMoa1414428. Epub 2015 Apr 20. PMID 25891304
- [Background] Sledzinska A, Menger L, Bergerhoff K, Peggs KS, Quezada SA. Negative immune checkpoints on T lymphocytes and their relevance to cancer immunotherapy. Mol Oncol. 2015 Dec;9(10):1936-65. doi: 10.1016/j.molonc.2015.10.008. Epub 2015 Oct 26. PMID 26578451
- [Background] 14. Antonia SJ, Bendell JC, Taylor MH. Phase I/II study of nivolumab with or without ipilimumab for treatment of recurrent small cell lung cancer (SCLC): CA209-032. ASCO Annual Meeting. 2015.
- [Background] Taur Y, Jenq RR, Ubeda C, van den Brink M, Pamer EG. Role of intestinal microbiota in transplantation outcomes. Best Pract Res Clin Haematol. 2015 Jun-Sep;28(2-3):155-61. doi: 10.1016/j.beha.2015.10.013. Epub 2015 Oct 22. PMID 26590773
- [Background] Iida N, Dzutsev A, Stewart CA, Smith L, Bouladoux N, Weingarten RA, Molina DA, Salcedo R, Back T, Cramer S, Dai RM, Kiu H, Cardone M, Naik S, Patri AK, Wang E, Marincola FM, Frank KM, Belkaid Y, Trinchieri G, Goldszmid RS. Commensal bacteria control cancer response to therapy by modulating the tumor microenvironment. Science. 2013 Nov 22;342(6161):967-70. doi: 10.1126/science.1240527. PMID 24264989
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Xia Y, Medeiros LJ, Young KH. Immune checkpoint blockade: Releasing the brake towards hematological malignancies. Blood Rev. 2016 May;30(3):189-200. doi: 10.1016/j.blre.2015.11.003. Epub 2015 Nov 25. PMID 26699946
- [Background] Chinai JM, Janakiram M, Chen F, Chen W, Kaplan M, Zang X. New immunotherapies targeting the PD-1 pathway. Trends Pharmacol Sci. 2015 Sep;36(9):587-95. doi: 10.1016/j.tips.2015.06.005. Epub 2015 Jul 7. PMID 26162965
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Nishimura H, Nose M, Hiai H, Minato N, Honjo T. Development of lupus-like autoimmune diseases by disruption of the PD-1 gene encoding an ITIM motif-carrying immunoreceptor. Immunity. 1999 Aug;11(2):141-51. doi: 10.1016/s1074-7613(00)80089-8. PMID 10485649
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Xu F, Xu L, Wang Q, An G, Feng G, Liu F. Clinicopathological and prognostic value of programmed death ligand-1 (PD-L1) in renal cell carcinoma: a meta-analysis. Int J Clin Exp Med. 2015 Sep 15;8(9):14595-603. eCollection 2015. PMID 26628942
- [Background] Massi D, Brusa D, Merelli B, Falcone C, Xue G, Carobbio A, Nassini R, Baroni G, Tamborini E, Cattaneo L, Audrito V, Deaglio S, Mandala M. The status of PD-L1 and tumor-infiltrating immune cells predict resistance and poor prognosis in BRAFi-treated melanoma patients harboring mutant BRAFV600. Ann Oncol. 2015 Sep;26(9):1980-1987. doi: 10.1093/annonc/mdv255. Epub 2015 Jun 2. PMID 26037795
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] 29. Hodi FS, Sznol M, Kluger HM, McDermott DF, Carvajal RD, Lawrence DP. Long-term survival of ipilimumab-naive patients (pts) with advanced melanoma (MEL) treated with nivolumab (anti-PD-1, BMS-936558, ONO-4538) in a phase I trial. Journal of clinical oncology : official journal of the American Society of Clinical Oncology. 2014;32(Supplement):9002.
- [Background] McKinstry KK, Strutt TM, Swain SL. Regulation of CD4+ T-cell contraction during pathogen challenge. Immunol Rev. 2010 Jul;236:110-24. doi: 10.1111/j.1600-065X.2010.00921.x. PMID 20636812
- [Background] Ansell SM, Hurvitz SA, Koenig PA, LaPlant BR, Kabat BF, Fernando D, Habermann TM, Inwards DJ, Verma M, Yamada R, Erlichman C, Lowy I, Timmerman JM. Phase I study of ipilimumab, an anti-CTLA-4 monoclonal antibody, in patients with relapsed and refractory B-cell non-Hodgkin lymphoma. Clin Cancer Res. 2009 Oct 15;15(20):6446-53. doi: 10.1158/1078-0432.CCR-09-1339. Epub 2009 Oct 6. PMID 19808874
- [Background] Bashey A, Medina B, Corringham S, Pasek M, Carrier E, Vrooman L, Lowy I, Solomon SR, Morris LE, Holland HK, Mason JR, Alyea EP, Soiffer RJ, Ball ED. CTLA4 blockade with ipilimumab to treat relapse of malignancy after allogeneic hematopoietic cell transplantation. Blood. 2009 Feb 12;113(7):1581-8. doi: 10.1182/blood-2008-07-168468. Epub 2008 Oct 30. PMID 18974373
- [Background] Yu P, Steel JC, Zhang M, Morris JC, Waldmann TA. Simultaneous blockade of multiple immune system inhibitory checkpoints enhances antitumor activity mediated by interleukin-15 in a murine metastatic colon carcinoma model. Clin Cancer Res. 2010 Dec 15;16(24):6019-28. doi: 10.1158/1078-0432.CCR-10-1966. Epub 2010 Oct 5. PMID 20924130
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] 35. Blazer BR, O'Connor RS, Milone MC, et al. Role of PD-1/PD-l1 in Acute and Chronic Graft Versus Host Disease. Blood: 126: (23).
- [Background] 36. Davids MS, Haesook TK, Costello CL, et al. A Multicenter Phase I/Ib Study of Ipilimumab for Relapsed Hematologic Malignancies after Allogeneic Hematopoietic Stem Cell Transplantation. Blood: 126 (23).
- [Background] 37. Herbaux C, Gauthier J, Brice P. Nivolumab Is Effective and Reasonably Safe in Relapsed or Refractory Hodgkin's Lymphoma after Allogeneic Hematopoietic Cell Transplantation: A Study from the Lysa and SFGM-TC.